CLINICAL TRIAL: NCT00464074
Title: Multi-center, Open-Label Study to Evaluate the Effects of Natalizumab Treatment on Fatigue and Cognition in Subjects With Relapsing Forms of MS
Brief Title: Evaluation of Natalizumab for thE Relief of MS Associated FatiGue
Acronym: ENER-G
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 001-06-NAT
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Multiple Sclerosis
Keywords: fatigue; Tysabri; cognition
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to study the effects of TYSABRI® treatment on fatigue and cognition in patients with relapsing forms of MS.

DETAILED DESCRIPTION:
TYSABRI® treatment has already demonstrated significant improvement in the quality of life (QoL) of patients with MS. In particular, TYSABRI® add-on treatment to interferon beta-1a has demonstrated improvement in fatigue as measured by the Modified Fatigue Impact Scale (MFIS). Both patients and neurologists report that patients have experienced significant improvements in fatigue shortly after initiating TYSABRI® treatment. Fatigue is both a common and a disabling symptom of MS. Further, there is evidence that fatigue contributes to cognitive difficulties in patients with MS. This study aims to study the effects of TYSABRI® treatment on fatigue and cognition in patients with relapsing forms of MS.

The primary objective of this study is to determine the effects of TYSABRI® treatment on fatigue in subjects with relapsing forms of MS as measured by changes in patient-reported Visual Analog Scale for Fatigue (VAS-F).

Primary endpoint is the change in the following:

1. Visual Analog Scale for Fatigue (VAS-F) at three months after initiating treatment with TYSABRI®.

Secondary objectives are to measure changes in patient-reported Modified Fatigue Impact Scale (MFIS) and Fatigue Severity Scale (FSS).

Secondary endpoints are changes in the following:

1. Modified Fatigue Impact Scale (MFIS)
2. Fatigue Severity Scale (FSS)

The tertiary objective of this study is to explore for any effects of TYSABRI® treatment on cognition by assessing changes in the Automated Neuropsychology Assessment Metrics (ANAM).

Tertiary endpoints are changes in the Automated Neuropsychology Assessment Metrics (ANAM) consisting of:

* Traditional Continuous Performance Test
* Running Memory Continuous Performance Test
* Simple Response Time
* Procedural Response Time
* Coding Substitution
* Mathematics
* Logical Relations
* Matching-to-Sample
* Stanford Sleepiness Scale

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of relapsing forms of MS.
2. Patients having an inadequate response to or unable to tolerate alternate MS therapies.
3. Patient must be enrolled in the TOUCH prescribing program.
4. Recent MRI as part of the TOUCH prescribing program.
5. Patient must be between 18 and 55 years of age, inclusive.
6. EDSS between 0 and 5.5, inclusive.
7. Able to provide written informed consent.
8. Capable of completing the fatigue (MFIS, FSS, and VAS-F) and cognition (ANAM) sessions.
9. A baseline VAS-F average score of > 60.
10. Patient must be naÃƒ-ve to TYSABRI® treatment.

Exclusion Criteria:

1. Patients not enrolled in the TOUCH prescribing program.
2. History or presence of progressive multifocal leukoencephalopathy (PML).
3. Diagnosis of primary progressive MS (PPMS) or secondary progressive MS (SPMS) without relapses.
4. Immunocompromised in the judgment of the investigator.
5. Allergy or hypersensitivity to TYSABRI®.
6. Prior history or current presence of a clinically significant medical illness or laboratory abnormality, including any significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric, renal, and/or other major disease, that, in the opinion of the investigator, would preclude the administration of TYSABRI®.
7. Women pregnant, breast feeding, or planning to become pregnant and women who are not postmenopausal or surgically sterile, and unwilling to practice contraception.
8. A baseline average VAS-F score of < 60.
9. Problems with upper extremity dexterity that could preclude usage of a computer mouse.
10. With educational completion below 8th grade school equivalent or non-fluent in English.
11. Any other reason, in the opinion of both the Investigator and/or Sponsor, the patient is determined not suitable for study participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: multicenter clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2010-07-31 (Actual); Study Completion 2010-07-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for Fatigue (VAS-F) | at three months after initiating treatment with TYSABRI®

CONTACTS AND LOCATIONS:
Locations (29):
- United States (28):
  - Research Site, Phoenix, Arizona
  - Research Site, Fresno, California
  - Research Site, Atlanta, Georgia
  - Research Site, Idaho Falls, Idaho
  - Research Site, Evanston, Illinois
  - Research Site, Lake Barrington, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, West Des Moines, Iowa
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Boston, Massachusetts
  - Research Site, Lexington, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Patchogue, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Anderson, South Carolina
  - Research Site, Franklin, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Salt Lake City, Utah
  - Research Site, Seattle, Washington
  - Research Site, Charleston, West Virginia
  - Research Site, Waukesha, Wisconsin
- Research Site, Guaynabo, Puerto Rico